CLINICAL TRIAL: NCT05262738
Title: Misoprostol Dosing in BMI Greater Than 30: A Randomized Controlled Trial
Brief Title: Misoprostol Dosing in BMI Greater Than 30
Acronym: MD30 RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lorie Harper, Maternal Fetal Medicine Division Director, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002350
Record Dates: First submitted 2022-01-25; First posted 2022-03-02 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy Related; Obesity; Labor Onset and Length Abnormalities
Keywords: Induction of Labor; Cervical Ripening; Misoprostol; Obesity
MeSH Terms: conditions — Obesity | interventions — Methods; Misoprostol

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups (intervention versus control) in parallel for the duration of the study. Randomization will occur according to a predetermined computer-generated stratified randomization scheme prepared by a study statistician.
Who Masked: Participant, Care Provider
Masking Description: This study will be double blinded with the research participants and providers/nursing masked to the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 50 Micrograms Vaginal Misoprostol (Intervention) (Experimental): Subjects in this arm will be randomized to the 50 micrograms of vaginal misoprostol (intervention) group, they will be admitted to labor and delivery and undergo placement of 50 micrograms of intravaginal misoprostol every 4 hours for cervical ripening.
  Interventions: Drug: 50 Micrograms Vaginal Misoprostol (Intervention)
- 25 Micrograms Vaginal Misoprostol (Control) (Active Comparator): Subjects in this arm will be randomized to the 25 micrograms of vaginal misoprostol (control) group, they will be admitted to labor and delivery and undergo placement of 25 micrograms of intravaginal misoprostol every 4 hours for cervical ripening.
  Interventions: Drug: 25 Micrograms Vaginal Misoprostol (Control)

INTERVENTIONS:
Drug: 50 Micrograms Vaginal Misoprostol (Intervention) — Subjects will undergo cervical ripening with 50 micrograms of vaginal misoprostol every 4 hours.
  Other Names: Cytotec
  Arms: 50 Micrograms Vaginal Misoprostol (Intervention)
Drug: 25 Micrograms Vaginal Misoprostol (Control) — Subjects will undergo cervical ripening with 25 micrograms of vaginal misoprostol every 4 hours.
  Other Names: Cytotec
  Arms: 25 Micrograms Vaginal Misoprostol (Control)

SUMMARY:
The investigators are performing a randomized controlled-trial investigating if 50mcg (compared to 25 mcg) of vaginal misoprostol reduces the time from induction start to delivery in obese women.

DETAILED DESCRIPTION:
As of 2019, almost 1 in 4 women in the United States had their labor induced with almost 9 in 10 women requiring different methods to prepare their cervix for induction. There have been several research studies in the past designed to look at the fastest and safest method for labor induction, however very few studies have been done in women with a Body Mass Index (BMI) greater than or equal to 30 kg/m2.

Women with a BMI greater than or equal to 30 kg/m2, also classified as Obesity, are known to have longer labor induction times and experience more "failed" labor inductions requiring cesarean delivery (C-Sections). Obese women are also at a higher risk of developing complications during labor and postpartum such as excessive vaginal bleeding and infections.

Due to limited information, the American College of Obstetricians and Gynecologists (ACOG) currently recommends a standard dosing of 25 or 50 micrograms of vaginal misoprostol for labor induction in all women. However, there are studies which specifically compared the 25 microgram and 50 microgram misoprostol doses and found that women have significantly shorter time to deliveries without any harmful effects to mother or baby.

The investigators will conduct a randomized controlled trial to determine if 50 micrograms of vaginal misoprostol, when compared to the standard 25 micrograms, reduces the time from the start of labor induction to delivery in obese women. Women who are admitted to Labor & Delivery for the purposes of labor induction will be randomized to undergo either 25 micrograms or 50 micrograms of vaginal misoprostol for cervical ripening. Women and their infants will be followed until the time of their discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation
2. Age 18 years or older
3. Gestational age >= 36 weeks
4. BMI >= 30 kg/m2 at time of labor induction
5. Cephalic presentation (including successful external cephalic version)
6. Cervical dilation <= 3cm
7. Intent to proceed with cervical ripening

Exclusion Criteria:

1. Contraindication to vaginal delivery (placenta previa, vasa previa, prior classical cesarean, non-vertex presentation, etc.)
2. Contraindication to prostaglandin administration (significant allergy, prior cesarean delivery, etc.)
3. Multiple gestations
4. Gestational age < 36 weeks
5. Non-reassuring fetal heart tracing
6. Evidence of clinical chorioamnionitis
7. Significant vaginal bleeding with concern for abruption
8. Prior cesarean delivery or uterine surgery
9. Major fetal anomaly or demise
10. Cervix >3cm
11. No intention to proceed with cervical ripening (not indicated, favorable bishop score, plan for Oxytocin administration, etc.)
12. Uterine tachysystole (defined as >= 5 contractions within a 10m period)
13. Fetal Growth Restriction (EFW <= 5% or elevated/absent/reversed Umbilical Artery dopplers)
14. Inability to give consent (inability to read/write in English or Spanish)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorie Harper, MD, MSCI, Study Director — Division Chief, Maternal-Fetal Medicine
Locations (1):
- University of Texas at Austin Dell Medical School, Department of Women's Health, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] McDonagh M, Skelly AC, Tilden E, Brodt ED, Dana T, Hart E, Kantner SN, Fu R, Hermesch AC. Outpatient Cervical Ripening: A Systematic Review and Meta-analysis. Obstet Gynecol. 2021 Jun 1;137(6):1091-1101. doi: 10.1097/AOG.0000000000004382. PMID 33752219
- [Background] Carbone JF, Tuuli MG, Fogertey PJ, Roehl KA, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):247-252. doi: 10.1097/AOG.0b013e31827e5dca. PMID 23303106
- [Background] Viteri OA, Tabsh KK, Alrais MA, Salazar XC, Lopez JM, Fok RY, Chauhan SP, Sibai BM. Transcervical Foley Balloon Plus Vaginal Misoprostol versus Vaginal Misoprostol Alone for Cervical Ripening in Nulliparous Obese Women: A Multicenter, Randomized, Comparative-Effectiveness Trial. Am J Perinatol. 2021 Aug;38(S 01):e123-e128. doi: 10.1055/s-0040-1708805. Epub 2020 Apr 16. PMID 32299108
- [Background] Al-Ibraheemi Z, Brustman L, Bimson BE, Porat N, Rosenn B. Misoprostol With Foley Bulb Compared With Misoprostol Alone for Cervical Ripening: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):23-29. doi: 10.1097/AOG.0000000000002403. PMID 29215514
- [Background] Adhikari EH, Nelson DB, McIntire DD, Leveno KJ. Foley Bulb Added to an Oral Misoprostol Induction Protocol: A Cluster Randomized Trial. Obstet Gynecol. 2020 Nov;136(5):953-961. doi: 10.1097/AOG.0000000000004123. PMID 33030881
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK. Births: Final Data for 2019. Natl Vital Stat Rep. 2021 Apr;70(2):1-51. PMID 33814033
- [Background] Obesity. In: Cunningham F, Leveno KJ, Bloom SL, Dashe JS, Hoffman BL, Casey BM, Spong CY. eds. Williams Obstetrics, 25e. McGraw Hill; 2018.
- [Background] Rossi RM, Requarth EW, Warshak CR, Dufendach K, Hall ES, DeFranco EA. Predictive Model for Failed Induction of Labor Among Obese Women. Obstet Gynecol. 2019 Sep;134(3):485-493. doi: 10.1097/AOG.0000000000003377. PMID 31403588
- [Background] Knutson, Karin Britta MD; Leung, Katherine MPH; Allocco, Elizabeth Rose MD; Minor, Kathleen MD; Delpapa, Ellen MD; Lauring, Julianne MD Time to Delivery Following Induction of Labor in Obese Versus Normal-Weight Women [11S], Obstetrics & Gynecology: May 2019 - Volume 133 - Issue - p 205S
- [Background] Staudenmaier, Emily K. DO; Chatterton, Carolyn G. DO, MPH; Montanez, Marelli DO; Sampino, Isabella; Vullo, John J. DO; Gurram, Padmalatha MD, MSCTR Induction of Labor Compared With Expectant Management and Risk of Cesarean Delivery in Obese Women [7F], Obstetrics & Gynecology: May 2019 - Volume 133 - Issue - p 63S-64S
- [Background] Pevzner L, Powers BL, Rayburn WF, Rumney P, Wing DA. Effects of maternal obesity on duration and outcomes of prostaglandin cervical ripening and labor induction. Obstet Gynecol. 2009 Dec;114(6):1315-1321. doi: 10.1097/AOG.0b013e3181bfb39f. PMID 19935035
- [Background] Ellis JA, Brown CM, Barger B, Carlson NS. Influence of Maternal Obesity on Labor Induction: A Systematic Review and Meta-Analysis. J Midwifery Womens Health. 2019 Jan;64(1):55-67. doi: 10.1111/jmwh.12935. Epub 2019 Jan 16. PMID 30648804
- [Background] Wolfe KB, Rossi RA, Warshak CR. The effect of maternal obesity on the rate of failed induction of labor. Am J Obstet Gynecol. 2011 Aug;205(2):128.e1-7. doi: 10.1016/j.ajog.2011.03.051. Epub 2011 Apr 8. PMID 21621187
- [Background] Grobman WA, Bailit J, Lai Y, Reddy UM, Wapner RJ, Varner MW, Thorp JM Jr, Leveno KJ, Caritis SN, Prasad M, Tita ATN, Saade G, Sorokin Y, Rouse DJ, Blackwell SC, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Defining failed induction of labor. Am J Obstet Gynecol. 2018 Jan;218(1):122.e1-122.e8. doi: 10.1016/j.ajog.2017.11.556. Epub 2017 Nov 11. PMID 29138035
- [Background] Norman SM, Tuuli MG, Odibo AO, Caughey AB, Roehl KA, Cahill AG. The effects of obesity on the first stage of labor. Obstet Gynecol. 2012 Jul;120(1):130-5. doi: 10.1097/AOG.0b013e318259589c. PMID 22914401
- [Background] Stefely E, Warshak CR. Contraction frequency after administration of misoprostol in obese versus nonobese women. J Matern Fetal Neonatal Med. 2019 Nov;32(21):3526-3530. doi: 10.1080/14767058.2018.1465919. Epub 2018 Apr 30. PMID 29656680
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Sanchez-Ramos L, Kaunitz AM, Delke I. Labor induction with 25 microg versus 50 microg intravaginal misoprostol: a systematic review. Obstet Gynecol. 2002 Jan;99(1):145-51. doi: 10.1016/s0029-7844(01)01644-1. PMID 11777525
- [Background] Handal-Orefice RC, Friedman AM, Chouinard SM, Eke AC, Feinberg B, Politch J, Iverson RE, Yarrington CD. Oral or Vaginal Misoprostol for Labor Induction and Cesarean Delivery Risk. Obstet Gynecol. 2019 Jul;134(1):10-16. doi: 10.1097/AOG.0000000000003274. PMID 31188317
- [Background] Farah LA, Sanchez-Ramos L, Rosa C, Del Valle GO, Gaudier FL, Delke I, Kaunitz AM. Randomized trial of two doses of the prostaglandin E1 analog misoprostol for labor induction. Am J Obstet Gynecol. 1997 Aug;177(2):364-9; discussion 369-71. doi: 10.1016/s0002-9378(97)70199-6. PMID 9290452
- [Background] Diro M, Adra A, Gilles JM, Nassar A, Rodriguez A, Salamat SM, Beydoun SN, O'Sullivan MJ, Yasin SY, Burkett G. A double-blind randomized trial of two dose regimens of misoprostol for cervical ripening and labor induction. J Matern Fetal Med. 1999 May-Jun;8(3):114-8. doi: 10.1002/(SICI)1520-6661(199905/06)8:33.0.CO;2-5. PMID 10338065
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Lenoir-Wijnkoop I, van der Beek EM, Garssen J, Nuijten MJ, Uauy RD. Health economic modeling to assess short-term costs of maternal overweight, gestational diabetes, and related macrosomia - a pilot evaluation. Front Pharmacol. 2015 May 20;6:103. doi: 10.3389/fphar.2015.00103. eCollection 2015. PMID 26042038
- [Background] Harvey S, Rach D, Stainton MC, Jarrell J, Brant R. Evaluation of satisfaction with midwifery care. Midwifery. 2002 Dec;18(4):260-7. doi: 10.1054/midw.2002.0317. PMID 12473441
- [Derived] Saucedo AM, Alvarez M, Macones GA, Cahill AG, Harper LM. Optimal misoprostol dosing among patients with a body mass index greater than 30: a randomized controlled trial. Am J Obstet Gynecol. 2024 May;230(5):565.e1-565.e16. doi: 10.1016/j.ajog.2024.02.004. Epub 2024 Feb 15. PMID 38367750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Started | 92 | 88
Completed | 91 | 88
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control) | Total
Number analyzed (Participants) | 91 | 88 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.63 (7.48) | 27.49 (6.73) | 28.07 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 88 | 179
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 64 | 130
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 79 | 77 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Nulliparous [Count of Participants; unit: Participants] | 55 | 51 | 106

OUTCOME MEASURES:

1. Primary Outcome: Interval Time From Labor Induction Initiation to Delivery (Vaginal or Cesarean)
Time Frame: From baseline to the time of delivery (baseline is initiation of labor induction), up to 3 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
hours | 18.56 (9.92) | 21.59 (11.11)

2. Secondary Outcome: Interval Time From Labor Induction to Vaginal Delivery
Time Frame: From baseline (baseline is initiation of labor induction) to the time of vaginal delivery, up to 3 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
hours | 17.20 (9.22) | 19.00 (10.76)

3. Secondary Outcome: Number of Cesarean Deliveries
Time Frame: Assessed following delivery, through study completion which is estimated at 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 25 | 24

4. Secondary Outcome: Number of Participants Exhibiting Uterine Tachysystole
Description: Tachysystole is defined as greater than or equal to 5 contractions within a 10 minute period
Time Frame: Assessed 4 hours post-misoprostol placement
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 20 | 9

5. Secondary Outcome: Number of Participants Exhibiting Uterine Tachysystole With Fetal Decelerations
Description: Tachysystole is defined as greater than or equal to 5 contractions within a 10 minute period. Decelerations are defined by the 2008 NICHD Fetal Monitoring Terminology.
Time Frame: Assessed 4 hours post-misoprostol placement
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 2 | 2

6. Secondary Outcome: Number of Participants Receiving Terbutaline
Time Frame: From baseline to the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 2 | 1

7. Secondary Outcome: Number of Participants Diagnosed With Clinical Chorioamnionitis
Time Frame: From baseline to the time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 8 | 10

8. Secondary Outcome: Number of Participants Diagnosed With Postpartum Hemorrhage
Time Frame: Assessed at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
Participants | 12 | 17

9. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 1
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 1: Experience has shown that I can have appropriate and adequate control over my care.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 6 [6 to 7] | 6 [6 to 7]

10. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 2
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 2: The person(s) responsible for my care are/were caring and compassionate.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 7 [6 to 7] | 7 [6 to 7]

11. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 3
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 3: Problems that have arisen up to now have not been dealt with effectively.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 2 [1 to 4] | 2 [1 to 4]

12. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 4
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 4: My needs have been addressed with appropriate consideration for my time.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 6 [6 to 7] | 7 [6 to 7]

13. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 5
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 5: The overall organization of my care has not been appropriate.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 2 [1 to 2] | 2 [1 to 2]

14. Secondary Outcome: Patient Satisfaction Six Simple Questions, Question 6
Description: Assessed through validated survey, Six Simple Questions. Adapted from Harvey S, Rach D, et al. Evaluation of satisfaction with midwifery care. 2002 Dec; 18(4):260-7.
  Question 6: I would choose the same type of care for my next pregnancy.
  1=strongly disagree, 4 = neutral, 7=strongly agree.
  Title: Six simple questions Definition: A survey to assess patient satisfaction during their cervical ripening and induction.
  Ranges: 1-7 Best score: 7 Worst score: 1
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 7 [6 to 7] | 6.5 [6 to 7]

15. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 1)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of misoprostol, and likeliness of recommending method of induction to a friend.
  Questions 1: Worst amount of pain experienced during labor. Scale 0-10. 0 = no pain, 10 = pain as bad as it could possibly be.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 10 patient satisfaction.
  Ranges: 0-10 Best score: 10 Worst score: 0
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 8 [5 to 9] | 8 [5 to 9]

16. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 2)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of misoprostol, and likeliness of recommending method of induction to a friend.
  Questions 2: Overall pain that you experienced during labor. Scale 0-10. 0 = no pain, 10 = pain as bad as it could possibly be.
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 10 patient satisfaction.
  Ranges: 0-10 Best score: 10 Worst score: 0
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 6 [5 to 9] | 6.5 [5 to 9]

17. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 3)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of misoprostol, and likeliness of recommending method of induction to a friend.
  Questions 3: Worst amount of pain you experienced following placement of the misoprostol
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 10 patient satisfaction.
  Ranges: 0-10 Best score: 10 Worst score: 0
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 5 [4 to 7] | 5 [3 to 7]

18. Secondary Outcome: Patient Satisfaction (Labor Pain Scale, Question 4)
Description: Assessed through a survey (Labor pain scale). Survey assesses worst amount of pain during labor, overall amount of pain, pain associated with placement of misoprostol, and likeliness of recommending method of induction to a friend.
  Questions 4: How likely are you to recommend your method of induction to a friend or family member? Please rate from 0 (strongly recommend) to 10 (strongly DO NOT recommend).
  Title: Likert scale for patient satisfaction. Definition: A survey to assess patient satisfaction and experience during their cervical ripening and induction using a Likert scale. This is a way to assess from 0 to 10 patient satisfaction.
  Ranges: 0-10 Best score: 0 Worst score: 10
Time Frame: Assessed postpartum day one following delivery, up to 5 days post-delivery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
Number analyzed (Participants) | 91 | 88
score on a scale | 2 [0 to 5] | 2 [1 to 5]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 week.
Description: Definitions do not differ
Arm/Group | 50 Micrograms Vaginal Misoprostol (Intervention) | 25 Micrograms Vaginal Misoprostol (Control)
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/91 | 5/88
Other Adverse Events (participants affected / at risk) | 18/91 | 23/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 Micrograms Vaginal Misoprostol (Intervention) (N=91) | 25 Micrograms Vaginal Misoprostol (Control) (N=88)
Maternal ICU admission (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — ICU transfer
Neonatal ICU Admission (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (4) — Neonatal ICU Transfer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 Micrograms Vaginal Misoprostol (Intervention) (N=91) | 25 Micrograms Vaginal Misoprostol (Control) (N=88)
postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 17 (17)
wound complication (Surgical and medical procedures) | 1 (1) | 0 (0)
clinical endometritis (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
pRBC transfusion (Blood and lymphatic system disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Results may not be generalizable to all women undergoing induction, safety cannot be inferred as the incidence of adverse outcomes was low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT05262738/Prot_SAP_000.pdf